CLINICAL TRIAL: NCT05937984
Title: Advanced Controlled Transcranial Magnetic Stimulation to Modulate Neuroplasticity and Alleviate Pain in Diabetic Neuropathy
Brief Title: Treatment for Painful Diabetic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16418
Record Dates: First submitted 2023-06-08; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Painful Diabetic Neuropathy
Keywords: controlled transcranial magnetic stimulation; painful diabetic neuropathy; pain; neuroplasticity
MeSH Terms: conditions — Diabetic Neuropathies; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cTMS (Active Comparator): Controlled Transcranial Magnetic Stimulation (cTMS) will be delivered at 10 Hz, 1500 pulses targeting the hand representation of the left primary motor cortex. cTMS delivery will require ~9 min to complete. This intervention will be performed approximately 5 days per week for 2 weeks. In addition, participants will experience their standard medical care.
  Interventions: Device: Active Controlled Transcranial Magnetic Stimulation (cTMS)
- Sham cTMS (Sham Comparator): Sham cTMS will be delivered at as a placebo control. It is important to note that from the participant perspective, the sham stimulation will feel and sound identical to active cTMS. This will be performed approximately 5 days per week for 2 weeks. In addition, participants will experience their standard medical care.
  Interventions: Device: Sham Controlled Transcranial Magnetic Stimulation (cTMS)

INTERVENTIONS:
Device: Active Controlled Transcranial Magnetic Stimulation (cTMS) — cTMS is a non-invasive, non-painful procedure used to relieve chronic pain and promote short-term changes. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. 1500 pulses will be delivered at 10 Hz stimulation. Stimulation will be delivered at 80% of the resting motor threshold obtained from the right APB muscle. The delivery of cTMS requires 9 minutes in total.
  Arms: Active cTMS
Device: Sham Controlled Transcranial Magnetic Stimulation (cTMS) — A sham coil will be utilized for the sham cTMS condition. It is important to note that from the participant perspective, the sham stimulation will feel and sound identical to active. The location and all other parameters of Sham cTMS will be identical to Active cTMS.
  Arms: Sham cTMS

SUMMARY:
Painful diabetic neuropathy (pDN) occurs in a subset of diabetic patients, and is characterize by burning, shooting, and electric shock-like pain in the arms and legs. This represents a major health crisis, given the increasing prevalence of pDN and the significant impact it has on quality of life. However, there is limited evidence of effective therapies for pDN pain relief. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive form of brain stimulation that may be a promising therapy for pDN. Previous research has shown that rTMS reduces neuropathic pain in pDN (1, 2, 3). While this is promising, it is important to note that rTMS is effective for ~50% of patients with neuropathic pain. (4, 5). Recent advancements in rTMS technology have created the opportunity for remarkable strides in the effectiveness of this potential therapy. This new development called controlled pulse parameter TMS (cTMS) increases the magnitude and longevity of TMS-induced effects. Although not tested in chronic pain, cTMS possess the power to make transformative changes in pDN, potentially yielding greater and widespread improvements in pain. The overarching goal of the proposed research is to assess the effects of a 5-day cTMS stimulation protocol on measures of pain and neurological function in individuals with pDN.

1. Kwak S, Choi SG, Chang GS, & Yang MC (2022). Short-term Effect of Repetitive Transcranial Magnetic Stimulation on Diabetic Peripheral Neuropathic Pain. Pain Physician, 25(2), E203-E209.
2. Abdelkader AA, Gohary AME, Mourad HS, & Salmawy DAE (2019). Repetitive tms in treatment of resistant diabetic neuropathic pain. Egyptian Journal of Neurology, Psychiatry and Neurosurgery, 55(1).
3. Onesti E et al. (2013). H-coil repetitive transcranial magnetic stimulation for pain relief in patients with diabetic neuropathy. European Journal of Pain (United Kingdom), 17(9).
4. Attal N et al. (2021). Repetitive transcranial magnetic stimulation for neuropathic pain: a randomized multicentre sham-controlled trial. Brain, 144(11).

65. Dongyang L et al. (2021). Posterior-superior insular deep transcranial magnetic stimulation alleviates peripheral neuropathic pain - A pilot double-blind, randomized cross-over study. Neurophysiologie Clinique, 51(4).

DETAILED DESCRIPTION:
Background: Diabetic neuropathy is one of the most common complications of diabetes occurring in ~50% of patients [1, 2]. Of these individuals, ~20% will develop painful diabetic neuropathy (pDN) [3] as a consequence of abnormal changes in the peripheral somatosensory system [4]. pDN is characterized by sensory changes including hyperalgesia, allodynia, paresthesia, and burning, shooting, and electric shock-like pain affecting lower and upper extremities [4-6]. pDN is a result of high glucose concentrations that damages peripheral nerves [7] resulting in hyperexcitability of nociceptive neurons in the dorsal horn and central sensitization [8]. pDN is also marked by alterations in the central nervous system [6] including the descending modulatory system [9] and maladaptive changes to somatosensory and motor areas [10]. pDN is associated with decreased quality of life, anxiety, and depression [5]. The treatment of pDN currently involves opioid agonist, antidepressants, and anticonvulsants however, these drugs are associated with undesired side effects [11] and only achieve a 50% reduction in pain with delayed onset [12]. Importantly, the prevalence of pDN is increasing [13] and given the limited effectiveness of pharmacological interventions, pDN represents a major healthcare crisis.

Repetitive transcranial magnetic stimulation (rTMS) may be a beneficial therapy for patients with pDN. Sham controlled studies [14-19] and meta-analyses [20-23] have demonstrated that high frequency rTMS stimulation applied to the primary motor cortex reduces symptoms of neuropathic pain in heterogenous groups of patients [24]. Our lab recently demonstrated that rTMS is effective at alleviating electric attacks in an individual with NP following SCI [25]. rTMS is also effective in pDN. Yang [26] found analgesic relief one day following stimulation to the hand representation of the primary motor cortex that persisted for 1 week. rTMS was also associated with significant improvements in physical and mental health measured using the SF-36 physical component score and mental component score respectively [26]. Abdelkader [27] indicated pain relief at 3 weeks post rTMS in patients with insulin-dependent and non-insulin-dependent pDN as well as improvements in lower limb nerve conduction latency and velocity. Comparatively, Onesti [8] targeted the leg representation in the primary motor cortex. rTMS reduced pain compared to sham immediately post stimulation but did not persist at three weeks [8]. rTMS also produced a depression of spinal nociceptive neurons as indicated through a decrease in the area of nociceptive flexion RIII reflex [8]. This finding suggests that rTMS increases the firing rates of cells in motor cortex and increases corticospinal excitability and neuroplasticity. These changes are thought to modulate descending inhibitory pain pathways through spinal interneural networks producing hypoexcitability of spinal nociceptive neurons [8]. Although the few studies in pDN demonstrate promise, it is important to note that rTMS is effective for ~50% of patients with neuropathic pain [24, 28] leaving much room for further improvement.

Recent advancements in rTMS technology have created the opportunity for remarkable strides in neuroplasticity. This new development called controlled pulse parameter TMS (cTMS) increases the magnitude and longevity of rTMS induced plasticity in humans [29, 30]. Fundamental to previous (i.e. traditional) rTMS is the biphasic pulse shape that are used during stimulation. In cTMS, pulses are monophasic and modifiable, and can be delivered at high rates used in rTMS [31, 32]. Although not tested in chronic pain, cTMS possess the power to make transformative changes in pDN, potentially yielding greater and widespread improvements in pain. The overarching goal of the proposed research is to assess the effects of a 10-day cTMS stimulation protocol on measures of pain, neuroplasticity, and somatosensory function in individuals with pDN.

How is cTMS thought to induce neuroplasticity and reduce pain? The primary motor cortex (M1) is directly implicated in modulating pain signals [33] through descending inhibitory control to thalamus [34, 35] and its connections with pain processing areas [36] including somatosensory [37] anterior cingulate cortex and prefrontal cortices [38, 39]. The analgesic effect of rTMS is suggested to occur by re-establishing both intracortical inhibition [40], GABAergic inhibition [41, 43], and descending inhibitory control [34, 35]. cTMS may more readily activate and cause change in the circuits projecting to these areas. Specifically, monophasic pulses delivered with repetitive cTMS produce larger and more long-lasting changes in cortical excitability [29] and greater depths of inhibition compared to traditional biphasic rTMS [30]. Monophasic pulses also produce more reliable cortical responses in cortical excitability, intracortical and GABAergic inhibition [44]. These findings have been suggested to occur as a result of the uniform pattern of cortical activation from monophasic pulses. Monophasic pulses produce greater global mean field power (GMFP) measured through electroencephalography (EEG) compared to biphasic [31]. Specifically, biphasic pulses may activate populations of both excitatory and inhibitory neurons which may dampen the overall effects of the stimulation protocol [29]. Taken together, cTMS may facilitate a greater propensity for change in these circuits and ultimately pain relief when applied to individuals with NP. The specific aims of this study in pDN are to:

1. Investigate the effects of a 10-day cTMS intervention on pain symptoms. The investigators hypothesize that cTMS will produce analgesic relief that will be associated with changes in neuroplasticity and somatosensory function compared to sham. Importantly, the effect of real and sham cTMS will be explored within individuals.
2. To explore the feasibility of the 10-day cTMS intervention. This will inform the utility of cTMS interventions in future treatments studies. In addition, the patient perceived change from the intervention will be assessed to improve the patient experience for future studies.
3. To assess the effects of the 10-day cTMS intervention on neurophysiology and somatosensory function. It is hypothesized that cTMS will produce neuromodulatory effects associated with increased cortical excitability, GABAergic inhibition, neuroplasticity, and improve somatosensory function compared to sham.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of painful diabetic neuropathy (pDN)

Exclusion Criteria:

* a known history of moderate to severe chronic pain other than pDN
* daily use of opioids prior to the pDN diagnosis
* contraindications to TMS
* known psychological diagnosis affecting comprehension and inability to participate in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS-29 v2.0 Profile | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  Using numerical rating (0 to 5) to assess the change in seven health domains including physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles and activities, and pain interference. Each category consists of 4 questions. Also uses a numerical rating to asses pain intensity (0-10).

SECONDARY OUTCOMES:
Number of responders to active cTMS | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  Defined as participants who experienced a reduction in NRS of at least 2 points at T1 or T4
Change in Patient Perceived Global Index of Change (PGIC) | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  1-7 Likert Scale: Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse.
Change in Pain catastrophizing scale-EN-SF | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  Will be used to assess the patients feeling and emotion related to their pain experience
Compliance of treatment sessions | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  Compliance of sessions is defined as a minimum of attending 3 sessions per week for 2 weeks.
Change in neurophysiological assessment | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  This will include assessments of Motor-evoked potentials (MEPs), short-intracortical inhibition (SICI), contralateral silent period (cSP) and motor maps obtained with single-pulse TMS (note: this form of TMS does not induce neuroplasticity like cTMS, but is instead used to assess the baseline excitability of the primary motor cortex)
Change in quantitative sensory testing | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  Will be used in this study to assess somatosensory function to determine underlying pain mechanisms for pain phenotypes. QST will be used to measure detection thresholds for cold, warm, vibration, and mechanical stimuli. Pain thresholds will be assessed for cold, heat, mechanical, and pressure stimuli. In addition, allodynia will be measured.
Change in nerve conduction assessments | Day 1 of intervention, 24 hours post intervention, and 1 week post intervention
  Nerve conduction measures will be acquired from bilateral upper and lower limbs. These will include both motor (tibial and ulnar) and sensory nerves (superficial peroneal, sural, and ulnar). Nerve conduction outcomes will include latencies, amplitudes, and conduction velocities and F-waves for the aforementioned nerves. In addition to nerve conduction, participants with lower limb pDN will have Hoffman-reflex assessments performed on bilateral lower limb. For all participants, the maximum M-wave (M-Max) of the right APB muscle will be acquired.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada